CLINICAL TRIAL: NCT02084147
Title: PET-MRI: Evaluation, Optimization and Clinical Implementation
Brief Title: PET-MRI in Diagnosing Patients With Cancer, Cardiac Diseases, or Neurologic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE16Z12; NCI-2014-00376 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE16Z12 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Disease; Dementia; Inflammatory Disease; Fever of Unknown Origin; Vasculitis; Osteomyelitis; FDG Avid Cancers
MeSH Terms: conditions — Heart Diseases; Dementia; Fever of Unknown Origin; Vasculitis; Osteomyelitis | interventions — Positron-Emission Tomography; Tomography, Emission-Computed; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET-CT and PET-MRI (Experimental): Patients undergo PET-CT over approximately 30 minutes and PET-MRI over approximately 45-90 minutes.
  Interventions: Device: positron emission tomography; Device: computed tomography; Device: magnetic resonance imaging

INTERVENTIONS:
Device: positron emission tomography — Undergo PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Device: computed tomography — Undergo CT
  Other Names: tomography, computed; CT
Device: magnetic resonance imaging — Undergo MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This randomized pilot clinical trial studies how well positron emission tomography (PET)-magnetic resonance imaging (MRI) works compared to standard-of-care PET-computed tomography (CT) in diagnosing patients with cancer, cardiac diseases, or neurologic diseases. PET-MRI combines two imaging methods that can be used to evaluate disease. PET-MRI is similar to standard-of-care PET-CT, but exposes the patient to less radiation. It is not yet known whether PET-MRI produces better image quality than PET-CT in diagnosing patients with cancer, cardiac disease, or neurologic disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess and optimize image quality of PET and MRI focusing on technical artifacts and their correction.

II. To assess the accuracy of PET quantification based on MR attenuation correction (MRAC) derived from various MRI sequences and reconstruction algorithms including the effect of routinely used Gadolinium-based contrast agents on MRAC.

III. To determine the clinical and diagnostic accuracy of PET-MRI in comparison to standard-of-care diagnostic imaging.

IV. To assess the efficacy and workflow in combining PET and MRI in one single examination as compared to separate imaging studies.

V. To assess the potential for radiation dose reduction if PET-CT is substituted by PET-MRI, thus avoiding the radiation exposure from the CT-component.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated PET/PET-CT (with or without clinically indicated diagnostic MRI)
* Presenting with one of the four conditions specified below

  * Fludeoxyglucose F 18 (FDG) avid cancers
  * Cardiac disease (cardiac viability assessment)
  * Neurologic disorders (dementia)
  * Inflammatory disease (for example fever of unknown origin, vasculitis, osteomyelitis)

Exclusion Criteria:

* Pregnancy and lactation
* Contraindications to undergo MRI
* Cardiac pacemaker and metal devices (as specified in a separate MRI Informed consent)
* Claustrophobia or inability to tolerate MRI examination (lay still for approximately 1 hour and hold breath intermittently)
* Previously known allergies against MRI contrast agents (exclusion criterion only for contrast enhanced MRI)
* Renal insufficiency: glomerular filtration rate (GFR) < 40ml/min/1.73m^2 and following European Society of Urogenital Radiology (ESUR) guidelines (exclusion criterion only for contrast enhanced MRI)
* Individuals who are not willing or capable of giving informed consent or assent (with legal guardian consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ros, MD, MPH, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET-CT and PET-MRI
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed study
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 72
Age, Customized [Count of Participants; unit: Participants]
  10-19 years | 4
  20-29 years | 1
  30-39 years | 3
  40-49 years | 4
  50-59 years | 25
  60-69 years | 17
  70-79 years | 14
  80-89 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 50
  More than one race | 8
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Overall Image Quality Scores
Description: Overall image quality scores obtained from the two imaging modalities will be compared with the hypothesis that hybrid PET-MRI images is as good as PET-CT images or superior (not inferior) to the PET-CT images. Evaluation of overall image quality will be assessed using the following criteria: 1=excellent, 2=good, 3=acceptable, 4=poor, 5=not acceptable. A Wilcoxon (Mann-Whitney) rank-sum test with a 0.100 significance level will be used.
Time Frame: Day 1
Population: No data was obtained from this study group as the patient cohort was inconsistent
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 0

2. Primary Outcome: Lesion Based Standard Uptake Values (SUV)
Description: Lesion based SUV will be estimated and compared for PET-MR and PET-CT images in normal organs and compared. A two-sided two-sample t-test will be used to show significance of difference.
Time Frame: Day 1
Population: No data was obtained from this study group as the patient cohort was inconsistent
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 0

3. Primary Outcome: Area Under the Receiver Operating Characteristic Curve
Description: A two-sided z-test will be used to detect the difference in the area under the curve showing the sensitivity, specificity, positive and negative predictive values as well as accuracy of diagnostic information.
Time Frame: Day 1
Population: No data was obtained from this study group as the patient cohort was inconsistent
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 0

4. Primary Outcome: Time Effort Associated With the PET-MRI Versus PET-CT With MRI
Description: Statistical difference in time between PET-MRI versus sequential approach for PET-CT plus MRI. Workflow with shortest timely efforts and sufficient diagnostic information will be established as routine procedure.
Time Frame: Day 1
Population: No data was obtained from this study group as the patient cohort was inconsistent
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 0

5. Primary Outcome: Radiation Dose Reduction With PET-MRI
Description: Dose measurements will be used to calculate effective radiation dose in each patient. Dose calculations of effective dose will be used to estimate dose savings in omitting the CT component of PET-CT. Statistical tests will use a 0.10 significance level and will be 2-sided
Time Frame: Day 1
Population: No data was obtained from this study group as the patient cohort was inconsistent
Arm/Group | PET-CT and PET-MRI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At time of scan
Arm/Group | PET-CT and PET-MRI
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

LIMITATIONS AND CAVEATS:
No data was obtained from this study group as the patient cohort was inconsistent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes